CLINICAL TRIAL: NCT07198646
Title: Evaluation of the Correlation of Ultrasound Measurements of Quadratus Femoris Muscle Thickness and Ischiofemoral Distance With MR Measurements in Patients Diagnosed With Ischiofemoral Impingement by MR Imaging and Clinical Examination.
Brief Title: Correlation of Ultrasound and MRI Measurements of Quadratus Femoris Thickness and Ischiofemoral Distance in Clinically and Radiologically Diagnosed Ischiofemoral Impingement
Acronym: MRI USG
Status: Completed | Type: Observational
Sponsor: Kutay Can ÇAMLICA (Other)
Responsible Party: Sponsor-Investigator, Kutay Can ÇAMLICA, Resident Physician, Department of Physical Medicine and Rehabilitation, Sisli Hamidiye Etfal Training and Research Hospital
Organization: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Other Study IDs: 4500
Record Dates: First submitted 2025-09-21; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2024-08

CONDITIONS: Hip Pain Chronic; Impingement Syndrome
Keywords: Ischiofemoral impingement, quadratus femoris compression, hip pain diagnosis, ultrasound-MRI correlation, cost-effective imaging in hip pathology.

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to evaluate the correlation between ultrasound measurements of quadratus femoris muscle thickness and ischiofemoral distance, as well as clinical parameters, with MRI measurements in patients diagnosed with ischiofemoral impingement (IFI) through MRI imaging and clinical examination. The main questions it aims to answer are: Is there a correlation between ultrasound and MRI measurements of quadratus femoris muscle thickness and ischiofemoral distance in patients with clinically and radiologically confirmed IFI? How do clinical parameters relate to ultrasound and MRI findings in these patients? What is the intra- and inter-rater reliability of ultrasound measurements for these parameters? Participants will undergo ultrasound measurement of quadratus femoris muscle thickness and ischiofemoral distance, assessment of clinical parameters related to ischiofemoral impingement, and measurements performed twice by two independent raters to assess intra- and inter-rater reliability. Researchers will compare ultrasound and MRI measurements as well as clinical parameters to determine if ultrasound can serve as a reliable and cost-effective alternative for diagnosing ischiofemoral impingement.

DETAILED DESCRIPTION:
Ischiofemoral impingement (IFI) was first described in 1977 by Karl A. Johnson, and his study is widely regarded as the first clinical definition of the syndrome. IFI is defined as an extra-articular hip impingement syndrome resulting from the narrowing of the space between the ischium and the lesser trochanter, leading to compression of the quadratus femoris muscle and surrounding soft tissues, thereby causing clinical symptoms.

IFI findings are associated with edema and irritation of the quadratus femoris muscle, as well as secondary atrophic fatty degeneration in chronic cases. The primary symptom is posterior and lateral hip pain, often exacerbated by physical activity. Due to the close anatomical relationship between the quadratus femoris muscle and the sciatic nerve, irritation of the nerve may lead to pain radiating anteriorly, to the posterior thigh, and distally to the knee.

The etiology of IFI is multifactorial, involving congenital anatomical variations, post-traumatic sequelae, postoperative changes following hip surgery, and primary hip joint pathologies. Additional factors, such as femoral anteversion, acetabular retroversion, and abductor or adductor insufficiencies, may also contribute to its pathogenesis. The exact prevalence of IFI remains unknown, but it has been reported to be more common in females than in males, with a female-to-male ratio of approximately 3:1. This higher incidence in females is attributed to gender differences in pelvic morphology and a narrower ischiofemoral space. While IFI typically affects middle-aged and older adults, it has been observed across a wide age range (30-70 years). Although IFI generally presents unilaterally, bilateral involvement has been reported in 25-40% of cases, with no consensus in the literature regarding side predominance. The diagnosis of IFI requires a combination of detailed patient history, physical examination, and imaging techniques. Clinical tests such as the long-stride walking test and the ischiofemoral impingement test play a significant role in diagnosis, while MRI is considered the gold-standard imaging modality for confirmation.

The present study aims to investigate the correlation between ultrasound measurements and MRI findings in patients diagnosed with IFI through MRI and clinical examination. Specifically, ultrasound measurements of quadratus femoris muscle thickness and ischiofemoral distance will be evaluated for their consistency with MRI findings. Additionally, clinical parameters related to IFI will be assessed to explore their association with imaging results. The primary objective of this study is to determine the feasibility of using ultrasound, a more cost-effective imaging method, as an alternative diagnostic tool for IFI. The hypothesis is that by establishing a reliable correlation between ultrasound and MRI findings, it may be possible to implement a lower-cost and more accessible diagnostic approach for this condition.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years and younger than 65 years.
2. Patients diagnosed by MRI
3. Those with a body mass index below 25 kg/m2
4. those with hip pain or positive physical examination tests

Exclusion Criteria:

1. Sciatic nerve damage detected on EMG
2. Patients with operative ischiofemoral decompression
3. Corticosteroid or any injection to the hip in the last 3 months
4. History of peripheral nerve damage
5. Femoroacetabular impingement
6. Pregnancy
7. Malignancy
8. Inflammatory pathologies: rheumatic, septic
9. Coxarthrosis-Kelgren-Lawrence grade 3-4
10. Those who have undergone hip arthroplasty/surgery
11. Causes of lumbar radiculopathy, spondylolisthesis
12. Patients with increased femoral anteversion - patients with increased hip internal rotation (Toe-in)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients older than 18 years and younger than 65 years.
  2. Patients diagnosed by MRI
  3. Those with a body mass index below 25 kg/m2
  4. those with hip pain or positive physical examination tests
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Correlation of ultrasonographic ischiofemoral space (IFS) and quadratus femoris muscle thickness with clinical and MRI parameters | Baseline (at enrollment)
  The primary outcome is to determine the relationship between ultrasonographically measured ischiofemoral space (IFS) and quadratus femoris muscle thickness with magnetic resonance imaging (MRI) findings (IFS and quadratus femoris space) and clinical parameters including pain intensity (Visual Analog Scale, VAS) and hip function (Harris Hip Score).

CONTACTS AND LOCATIONS:
Overall Officials: Jülide Öncü Alptekin, Professor, Study Director — Sisli Hamidiye Etfal Training and Research Hospital
Locations (1):
- Seyrantepe Hamidiye Etfal Training and Research Hospital, University of Health Sciences, Istanbul, Turkey, Istanbul, sarıyer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No